CLINICAL TRIAL: NCT00510289
Title: Phase II Trial of Sorafenib in Patients With Myelodysplastic Syndrome
Brief Title: Sorafenib in Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early closure of study due to poor response
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008151
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
Keywords: Sorafenib; Myelodysplastic Syndromes; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- all patients (Experimental): sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400 mg twice a day until progression or unacceptable toxicity develops.
  Other Names: Nexavar

SUMMARY:
The purpose of this study is to evaluate the efficacy of sorafenib in patients with Myelodysplastic Syndrome (MDS). Eligible subjects will receive Sorafenib administered at 400mg orally twice a day, given on days 1-28 of a 28-day cycle. Patients will be evaluated for hematological response after 2 cycles and then every 3 cycles thereafter for a maximum of 5 years from study entry. If a patient achieves a complete response they may receive an additional 6 cycles of therapy beyond documentation of complete response unless unacceptable toxicity occurs. For patients with partial response, hematological improvement or stable disease they will continue treatment until relapse, progression of disease, or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of primary or therapy-related myelodysplastic syndrome or myelodysplastic/ myeloproliferative disorders as defined by the WHO

  * Refractory anemia with excess blasts - 1 or 2
  * Chronic myelomonocytic leukemia type 2
  * Refractory anemia, refractory anemia with ringed sideroblasts, refractory cytopenia with multilineage dysplasia, refractory cytopenia with multilineage dysplasia with ringed sideroblasts, 5q- syndrome, myelodysplastic syndrome unclassified or chronic myelomonocytic leukemia type 1 if at least one of the following criteria is met: HgB < 10 g/dl, Platelets < 50,000/ul,ANC < 1,000 ul, Transfusion dependent defined as 2 transfusions within an 8 week period.
* Patients may have low, intermediate-1, intermediate-2 or high risk MDS or CMML.
* Patients are eligible without regard to prior treatment status except for allogenic bone marrow transplant.
* Patients must be 18 years of age or older.
* Patient has an estimated or measured creatinine clearance ≥30 ml/min at study enrollment.
* AST, ALT, total bilirubin ≤ than 2.5 times the upper limit of normal.
* ECOG performance status of 0-2.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control.
* Male subject agrees to use an acceptable method for contraception for the duration of the study therapy and for 2 weeks after study completion.

Exclusion Criteria:

* Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result within 2 weeks of enrollment. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs for this disease within 14 days of enrollment
* No growth factor support with erythropoietin, GCSF, or GMCSF within 28 days of enrolling in the study.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with another malignancy within the last one year (from documentation of remission) other than basal or squamous cell skin cancer or CIS of the cervix.
* Patients who underwent allogeneic stem cell transplant will be excluded.
* History of leukemia (having more than 20% blasts in blood or marrow)
* Current treatment with coumadin, heparin and its derivatives.
* Major surgery (including needle biopsy of visceral organs) for 1-month prior to study and fully recovered. In addition, no placement of a subcutaneous or tunneled venous access device for 3 days prior to study and adequately healed.
* Significant cardiac or vascular events within 6 months: acute MI, unstable angina, severe peripheral vascular disease (ischemic pain at rest class 3 or worse, non-healing ulcers/wounds, congestive heart failure (NHYA class ≥ 2), uncontrolled cardiac arrhythmias, and disseminated intravascular coagulation.
* No use of hematopoetic growth factors within 4 weeks of starting sorafenib.
* Known severe hypersensitivity to Sorafenib or any component of the formulation.
* Caution should be exercised with the concomitant use of other CYP3A4 inducers, such as rifampin, St. John's Wort, phenytoin, phenobarbital and dexamethasone.
* Uncontrolled hypertension with a systolic blood pressure greater than 160 or a diastolic blood pressure greater than 100 despite treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 years or older with an ECOG performance status of 0-2, and adequate renal and hepatic function with a diagnosis of primary or therapy-related MDS were eligible for this study. Patients were enrolled from 2006 to 2011 at Duke and Duke Oncology Network sites. The study was closed prematurely due to poor response and patient withdrawals.
Pre-assignment Details: Three patients were ineligible due to the presence of AML in the BM done at the time of screening.
Groups:
- All Patients: All patients who signed consent
Period: Overall Study
Arm/Group | All Patients
Started | 19 (All patients who consented)
Started Study Drug | 16 (3 patients progressed prior to starting study drug)
Completed | 7 (Completed at least one cycle of study drug and had disease assessments)
Not Completed | 12
Not completed — Withdrawal by Subject | 7
Not completed — Refused bone marrow biopsy | 2
Not completed — Lost to Follow-up | 1
Not completed — Progressed prior to starting drug | 2

BASELINE CHARACTERISTICS:
Population: All patients who signed consent
Arm/Group | All Patients
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Hematological Response
Description: Hematological response is defined as the number of subjects who achieve either a complete response (CR), Partial response (PR) or Hematologic improvement.(HI). HI is defined as peripheral blood counts with hemoglobin ≥11 g/dL, absolute neutrophil count ≥1x10(9)/L and platelet count ≥100x10(9)/L, and normal bone marrow morphology with no evidence of dysplasia or blasts. CR is defined as the disappearance of all signs and symptoms related to disease, along with HI. PR is defined as fulfilling the criteria for CR in the peripheral blood but blasts decreasing by 50% or more in the bone marrow or to a less advanced WHO classification pretreatment.
Time Frame: During treatment - up to a maximum of 5 years
Population: There were 16 subjects enrolled in the trial. 9 subjects refused further bone marrow biopsy to assess response to therapy. Therefore, there were 7 evaluable subjects. One subject experienced PR
Measure: Number; unit: participants
Groups:
- Evaluable Subjects: Patients who received at least one cycle of study drug and underwent bone marrow assessments
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 7
participants
  Partial Response | 1
  Complete Response | 0
  Hematologic Improvement | 0

2. Secondary Outcome: Number of Subjects Requiring Dose Reductions
Description: The number of subjects who took study drug for more than 1 cycle and required a dose reduction down to the next dose level.
Time Frame: While on study drug, a maximum of 5 years
Population: 7 Subjects completed beyond cycle 1. 4 of those subjects had dose reductions during the time they took study drug.
Measure: Number; unit: participants
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 7
participants | 4

3. Secondary Outcome: Time to Progression
Description: Time to progression will be defined as the number of months between on-study and the date of progression or death, whichever comes first, in subjects who took study drug for at least cycle 1.
Time Frame: 5 years
Population: 7 patients completed cycle one and had bone marrow biopsies to confirm response.
Measure: Median (Full Range); unit: months
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 7
months | 3.5 [2 to 7]

4. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the number of months from enrollment onto the study until death from any cause in subjects who took study drug for at least cycle 1.
Time Frame: 1 year from the last dose of study drug
Population: 7 subjects completed cycle 1 or beyond.
Measure: Mean (Full Range); unit: months
Groups:
- Evaluable Patients: Patients who received at least one cycle of study drug and underwent bone marrow assessments
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 7
months | 15 [5 to 40]

5. Secondary Outcome: Change in Microvessel Density
Description: Microvessel density will be measured before and after treatment, and the distribution of change across time will be summarized with descriptive statistics.
Time Frame: Measured before and after treatment
Population: This outcome was not analysed due to the early closure of the study.
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days after the last dose of study drug
Description: Serious Adverse Events/Other Adverse events are recorded whether or not they are thought to be related to the study drug. SAEs are listed for all patients who took at least one dose of study drug. Due to early study closure and patient withdrawals, Other AEs are listed for 9 patients only.
Groups:
- All Patients: SAEs are listed for all patients who took at least one dose of study drug. Due to early study closure and patient withdrawals, Other AEs are listed for 9 patients only.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=16)
Mucositis (Gastrointestinal disorders) | 1 (1)
Myositis (Infections and infestations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=9)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Ocular / Visual - Other (Eye disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI - Anus (Gastrointestinal disorders) | 1 (1)
Mucositis / stomatitis (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 (1)
Pain - Abdomen (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (11)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Pain - Chest / thorax NOS (General disorders) | 2 (2)
Pain - Other (General disorders) | 2 (3)
Rigors / chills (General disorders) | 1 (1)
Infection - Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC - Mucosa (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 (4)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 2 (3)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (1)
Metabolic / Laboratory - Other (Investigations) | 1 (1)
Platelets (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body / generalized (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal / Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (inflammation / damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 3 (4)
Neurology - Other (Nervous system disorders) | 1 (1)
Pain - Head / headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Mood Alteration - Anxiety (Psychiatric disorders) | 1 (1)
Mood Alteration - Depression (Psychiatric disorders) | 1 (1)
Renal / Genitourinary - Other (Renal and urinary disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hemorrhage, pulmonary / upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain - Throat / pharynx / larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Hair Loss / Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 3 (4)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The limitations of our study include the small sample size, the poor toxicity profile and the lack of response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes